CLINICAL TRIAL: NCT01812512
Title: Communication Skills Training for Heart Failure Self-Management in Telehealth
Brief Title: Telehealth Self Management for CHF
Acronym: TSM-CHF
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Never funded.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: William Jennings Bryan Dorn VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RRP 12-230
Record Dates: First submitted 2012-09-12; First posted 2013-03-18 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Heart Failure
Keywords: Heart Failure; Communication; Telemedicine; Veterans; Nurse-patient relations
MeSH Terms: conditions — Heart Failure; Communication | interventions — Educational Status; Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIPS for HF Intervention HT Training-Charleston-Pre/Post (Other): Group 1 (Charleston): In the proposed intervention, called Teaching for Interactive Patient Self-Management (TIPS) for Heart Failure (HF) , the observations from the previous RRP are used along with best practices from other studies of patient-centered communication in the VA , telephone coaching for chronic disease , problem-solving and counseling skills for telehealth nurse care managers , difficulties identified by patients working with the Health Buddy for telemonitoring , participation in provider-patient communication , essentials of patient education in heart failure process and content, and teach to goal theory to improve HF self-management for patients with low health literacy . Rather than an experimental trial, this implementation quasi-experimental pilot study examines pre- and post-training nurse practices and Veteran outcomes before and after communication skills training. The same intervention will then be delivered to Group 2 HT nurse care coordinators.
  Interventions: Behavioral: Teaching for Interactive Patient Self-Management (TIPS) for Heart Failure (HF
- TIPS for HF Intervention HT Training-Columbia-Pre/Post (Other): Group 2 (Columbia VAMC): To test the TIPS for HF educational intervention sufficiently in a sample not previously exposed to the information, the HT program at Dorn VA Medical Center in Columbia, South Carolina has volunteered to participate as a second study site. There are six nurse care coordinators who will be recruited; the larger number supports recruitment of a comparable number with 25 Veterans with HF to be recruited in the second site for a total of 50 Veterans. Both groups will use a purposeful sampling plan, beginning with an IRB-approved flyer for recruitment. The demographic make-up of the Charleston VAMC group is comparable Columbia HT group in age, race, and NYHA HF class. Also, consistent with an implementation quasi-experimental pilot study, the second site will examine pre-training and post-training nurse care coordinator communication practices and Veteran outcomes before and after communication skills training.
  Interventions: Behavioral: Teaching for Interactive Patient Self-Management (TIPS) for Heart Failure (HF

INTERVENTIONS:
Behavioral: Teaching for Interactive Patient Self-Management (TIPS) for Heart Failure (HF — The curriculum plan adapts components from the Rochester Participatory Decision-Making Scale (RPAD) and recent advances in communication skills training for chronic disease to develop a valid and reliable intervention specific to Home Telehealth (HT) shared decision making, effective telehealth communication, and patient self-management for heart failure (HF), using established best-practices and Veteran input. Veteran volunteers will participate in video recorded simulations to promote nurse care coordinator (NCC) active participation and problem-solving during the course. Scenarios are taken from transcribed actual HT interactions from the first exploratory RRP study of HT. The course is set up as one live session, one online module, and a final live session for more difficult conversations.

SUMMARY:
People with heart failure (HF) are hospitalized over a million times a year in the US at a cost over $39 billion dollars. About half of the patients are readmitted within 30 days. Despite a number of institutional reforms, cost and readmissions remain high in the VA. The VA Home Telehealth (HT) monitoring program decreases preventable readmissions, but HF readmissions remain increased in the VA. Despite an active and effective HT program, the Charleston VAMC has the highest HF readmission rate in VISN 7. Though the HT program introduces communication, self-management, and shared decision-making in initial training, previous QUERI RRP evaluation identified lower than expected levels of specific communication practices associated with the promotion of HF self-management and shared decision-making, mediated by the requirements of the technology.

DETAILED DESCRIPTION:
Clinical goals of the VA CHF QUERI identify best practices to empower Veterans and their caregivers for HF self-management. Recommendations of the American College of Cardiology/American Heart Association emphasize shared decision-making. In the previous preliminary study, coding of actual recordings of Veterans speaking with HT nurse care coordinators provided evidence of best practices and areas for improvement for intervention development. The effect of the HT technology as a mediator of Veteran-nurse communication requires particular re-framing in communication skills training to promote shared decision-making and self-management as recommended. This quasi-experimental study proposes the development of an evidence-based intervention to enhance HT training tailored for more effective communication for HF self-management and related outcomes.

Goals:

Phase 1 To conduct a pilot study as a quasi-experimental trial at two VAMC HT sites to determine acceptability, actual use, implementation, practicality, integration, potential for expansion, effect sizes and limited efficacy for an HT-specific communication skills intervention for HF Specific Aim 1.1a Development: Adapt components from the Rochester Participatory Decision-Making Scale (RPAD) and recent advances in communication skills training for chronic disease to develop a valid and reliable intervention specific to HT shared decision-making and telehealth communication using established best-practices and Veteran input; Specific Aim 1.1b Training/Implementation: Implement the developed intervention at two VAMCs; Specific Aim 1.2Booster: Introduce an audit and feedback loop of HF self-management outcomes for telehealth nurse practice as a booster to reinforce communication skills training.

Phase 2 To compare changes in Veteran outcomes after a telehealth communication skills intervention with documented previous practice for differences in: a) shared decision-making; b) Veteran perception of communication, education and self-management for HF, c) quality of life, and d) health service utilization and related costs before and after intervention Specific Aim 2.1: Formative Evaluation: Nurses: Conduct anonymous surveys of knowledge of HF and self-management strategies before and after training, qualitative interviews of reactions to the training course, and nurse care coordinator focus groups about the value of audit and feedback sessions after training.

Specific Aim 2.2: Formative Evaluation: Veterans - Phone record 25 Veterans with HF at two HT sites, for a total of 50 Veterans, speaking with nurse care coordinators before and after communication skills training followed by communication coding and discourse analysis.

Specific Aim 2.3: Summative Evaluation: Compare shared decision-making scores (SDM) measured by the RPAD, communication scores measured by the Four Habits Coding Scheme (FHCS), quality of life (Minnesota Living with Heart Failure Questionnaire), communication, education and self-management in HF as measured by the Improving Chronic Illness Care Evaluation (ICICE) scale, and patient HF hospitalization use (admissions and emergency) and with pre-training averages and with the post training averages at 1 and 3 months Rationale The technology of HT monitoring of Veterans with HF can inadvertently decrease participative communication consistent with shared decision-making and HF self-management. Application of communication skills training using evidence-based coach role competencies promises to improve Veteran engagement and participation in the VA Home Telehealth service with increased self-management and potential improvement in HF health service utilization. Improving engagement and participation in self-management should result in a quantifiably better Veteran quality of life, a reduction in hospital and ED admissions, and thus, a decrease in health care utilization costs for the VA.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic heart failure (CHF)
* enrollment in VA Home Telehealth (HT) program for at least 6 months
* Veteran who did not participate in the previous HT study

Exclusion Criteria:

* Veteran who is unable to communicate by telephone
* Veteran who does not pass the Clock Drawing Test for screening neurological problems at the initial visit

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Rochester Participatory Decision Making (RPAD) | pre and post (1 - 3 months)
  9 item scale that assess how the clinical issue was explained, discussion of uncertainties, clarification of agreement, identification of barriers, patients asked questions, medical language, physician validates open ended questions, checks for understanding

SECONDARY OUTCOMES:
Minnesota Living with Heart Failure Questionnaire | pre and post (1 - 3 months)
  To measure the effects of symptoms, functional limitations, psychological distress on an individual's quality of life, the MLHF questionnaire asks each person to indicate using a 6-point, zero to five, Likert scale how much each of 21 facets prevented them from living as they desired

CONTACTS AND LOCATIONS:
Overall Officials: Charlene A Pope, PhD MPH BSN, Principal Investigator — Ralph H. Johnson VA Medical Center
Locations (2):
- United States (2):
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC, Columbia, South Carolina